CLINICAL TRIAL: NCT03267147
Title: PREVALENCE OF ANTI-CYCLIC CITRULLINATED PEPTIDE (Anti-CCP) POSITIVITY AND SUBCLINICAL SIGNS OF INFLAMMATION IN PATIENTS WITH NEW ONSET OF NON-SPECIFIC MUSCULOSKELETAL SYMPTOMS POSSIBLY RELATED TO EARLY RHEUMATOID ARTHRITIS IN GENERAL PRACTICES IN GERMANY
Brief Title: PREVALENCE OF Anti-CCP POSITIVITY AND SUBCLINICAL SIGNS OF INFLAMMATION IN PATIENTS WITH NEW ONSET OF NON-SPECIFIC MUSCULOSKELETAL SYMPTOMS
Acronym: PANORA
Status: Completed | Type: Observational
Sponsor: Fraunhofer Institute for Translational Medicine and Pharmacology ITMP (Other)
Collaborators: Bristol-Myers Squibb (Industry); Goethe University (Other)
Responsible Party: Principal Investigator, Dr. Frank Behrens, Head of clinical research department, Fraunhofer Institute for Translational Medicine and Pharmacology ITMP
Other Study IDs: TMP-1016_01
Record Dates: First submitted 2017-07-04; First posted 2017-08-30 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Anti-CCP; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- antiCCP positive: Patients with a positive result in the anti-CCP quick test and positive in antiCCP ELISA will be examined by Rheumatologist for detection of RA symptoms and followed-up for 3 years or until RA diagnosis
  no intervention is given
  Interventions: Other: no intervention is given
- antiCCP negative: Patient with negative result in antiCCP quick test or negative antiCCP ELISA will be followed-up after one year (and 3 years for ELISA negative patients) with a short questionnaire if musculoskeletal symptoms are still present or if RA was diagnosed
  Interventions: Other: no intervention is given

INTERVENTIONS:
Other: no intervention is given — no intervention is given

SUMMARY:
Non-interventional, prospective, observational study to assess the relative risk of anti-CCP positive patients to develop (subclinical) signs of inflammation in accordance with early Rheumatoid Arthritis (RA) in a population without pre-classified RA but new1 onset of non-specific musculoskeletal (MSK) symptoms in general practices in Germany and subsequent 36 months follow-up by rheumatologists

DETAILED DESCRIPTION:
Studies of early arthritis cohorts have shown that a large number of early arthritis patients cannot be accurately diagnosed at their first visit, and hence are often referred as undifferentiated arthritis patients. If patients are found to be anti-CCP(+) when referred to the clinician, however, more than 90% develop RA within 3 years - in contrast to only 30% of the anti-CCP(-) patients. The presence of anti-CCP antibodies in undifferentiated arthritis therefore accurately predicts development of RA. Anti-CCP antibodies are very specific for RA, and they are produced at significant level very early in disease. The specificity of anti-CCP antibodies for the diagnosis of RA is high (94.1-99.0%). Moreover, it has been reported that anti-CCP antibodies can be present many years before the first visit to the clinic (up to 18 years). Furthermore, the presence of anti-CCP antibodies at the first visit to the clinician predicts radiographic progression, as demonstrated by many studies that have shown a strong association of anti-CCP positivity with the development of bone erosions.Early diagnosis of RA coupled with rational use of disease-modifying anti-rheumatic drugs (DMARD) has been shown to have a favourable effect on the course of the disease. Early and accurate diagnosis has therefore become increasingly important. Implementing anti-CCP quick tests in general practices could facilitate an early detection of RA or the allocation to a high risk RA group. This, in turn, would guarantee an early referral of the patient to a rheumatologist and together with other clinical examinations can aid in the early diagnosis and treatment. As has been shown in many studies an early intervention is vital to preserve joint function and to improve patient care. In this study, we want to assess the relative risk for patients derived from GPs in Germany with new onset of non-specific MSK symptoms and anti-CCP test positivity to develop (subclinical) signs of inflammation in accordance with early RA. Those patients will be identified in general practices and will be tested for anti-CCP status. Anti-CCP positive patients will then be introduced to a rheumatologist to validate anti-CCP status and examine presence of clinical signs of early RA in addition to subclinical signs of MSK inflammation. Furthermore, to focus on the possibility of early detection of anti-CCP before the onset of clinically active arthritis, patients will be followed-up by a rheumatologist until detection of early RA or up to 36 months in total. Early RA will be examined using standard of care for signs of inflammation including clinical examination for swollen and tender joints. In addition, ultrasound will be performed to assess joint inflammation as well as fluorescence optical imaging technique (Xiralite®) to sensitively illustrate changes in microvascularisation as a marker of subclinical inflammation. In cases of RA diagnosis, the study ends with the date of diagnosis and patients will receive treatment according to local guidelines earlier and medical care will be continued in clinical routine care conditions outside of the study. Moreover, the cooperation status between GPs and rheumatologists will be evaluated using qualitative interviews. Feasibility of the diagnosis of early RA in at risk patients as well as the feasibility of the transferral of these patients from the general practice to the rheumatologist will be assessed. Training of GPs for detection of early RA will be improved. Overall, the hypothesis of the study is that patients with new onset of unspecific MSK-symptoms and who are positive for anti-CCP, which both are risk factors for developing RA, will be earlier introduced to and monitored by a rheumatologist for proper clinical examination and potential treatment when establishing RA, which in turn will not only improve patient care, disease outcomes and quality of life, but might also be cost effective.

ELIGIBILITY:
Inclusion Criteria:

* New onset of non-specific MSK symptoms, including, but not limited to, arthralgia of the hands and the large joints such as wrists, knees, and shoulders
* Written informed consent obtained prior to the initiation of any study protocol-required procedures
* General understanding of study procedure and informed consent
* Age ≥ 18 and ≤ 65 years

Exclusion Criteria:

* RA diagnosed according to modified EULAR/ACR (american college of rheumatology)-criteria
* Other known arthritis
* Other known reasons for MSK symptoms, e.g. mechanical, traumatic, etc.
* MSK symptoms previously reported at another (general) practice
* Alcohol, drug or chemical abuse
* Underage or incapable patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: population without pre-classified RA but new onset of non-specific musculoskeletal (MSK) symptoms
Sampling Method: Non-Probability Sample
Enrollment: 986 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Determination of the relative risk in patients with new onset of non-specific MSK symptoms who are anti-CCP positive to develop (subclinical) signs of inflammation in accordance with early RA in general practices in Germany | every 6 months up to 3 years
  Determination if RA symptoms are present

SECONDARY OUTCOMES:
diagnosis of RA in the group of anti-CCP positive patients with new onset of non-specific MSK symptoms | every 6 months up to 3 years
subclinical signs of inflammation using routine examination methods in anti-CCP positive patients | every 6 months up to 3 years
subclinical signs of inflammation using fluorescence optical imaging technique in anti-CCP positive patients | every 6 months up to 3 years
subclinical signs of inflammation using ultrasound in anti-CCP positive patients | every 6 months up to 3 years
anti-CCP level over time in anti-CCP positive patients | over 3 years
EQ5D | every 6 months up to 3 years
  Questionnaire to assess Quality of Life profile of anti-CCP positive patients
SF36 | every 6 months up to 3 years
  Questionnaire to assess Quality of Life profile of anti-CCP positive patients
HAQ | every 6 months up to 3 years
  Questionnaire to assess disability profile of anti-CCP positive patients
PHQ-9 | every 6 months up to 3 years
  Questionnaire to assess depression profile of anti-CCP positive patients
WPAI | every 6 months up to 3 years
  Questionnaire to assess work ability profile of anti-CCP positive patients
assessment of time to disease in anti-CCP positive patients | every 6 months up to 3 years
assessment of correlation of anti-CCP level in anti-CCP positive patients | every 6 months up to 3 years
assessment quality of life (QoL) in anti-CCP positive patients | every 6 months up to 3 years
assessment work ability profile in anti-CCP positive patients | every 6 months up to 3 years
assessment subclinical signs of inflammation in anti-CCP positive patients | every 6 months up to 3 years
assessment risk of depression in anti-CCP positive patients | every 6 months up to 3 years
assessment of grade of disability in anti-CCP positive patients | every 6 months up to 3 years
diagnosis of RA in the group of ELISA test anti-CCP negative patients with new onset of non-specific MSK symptoms | 1 year
diagnosis of RA in the group of ELISA test anti-CCP negative patients with new onset of non-specific MSK symptoms | 3 years
diagnosis of RA in the group of quick test anti-CCP negative patients with new onset of non-specific MSK symptoms | 1 year
Qualitative assessment of general practitioners' (GP) routine care | 1 year
  qualitative interviews with the GP to evaluate current status of how patients with MSK symptoms are treated/forwarded in general practices

CONTACTS AND LOCATIONS:
Overall Officials: Frank Behrens, MD, Principal Investigator — Fraunhofer IME
Locations (1):
- CIRI, Frankfurt am Main, Hessia, Germany

IPD SHARING:
Plan to Share IPD: Undecided